CLINICAL TRIAL: NCT02579889
Title: Clinical Benefits of the Closed Loop Stimulation in Sinus Node Disease - B3 Study
Brief Title: Clinical Benefits of the Closed Loop Stimulation in Sinus Node Disease
Acronym: B3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopping criterion met (N. adjudicated EP1)
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA104
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sinus Node Disease
Keywords: Closed Loop Stimulation; Atrial Fibrillation; Stroke; Heart Failure; Pacemaker; ICD
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation; Stroke; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active group - CLS ON (Experimental): Device will be programmed in a dual-chamber DDD pacing mode with the Closed Loop Stimulation (CLS) function ON; Intervention: DDD+CLS
  Interventions: Device: DDD+CLS
- Control group - CLS OFF (Active Comparator): Device will be programmed in a dual-chamber DDD(R) pacing mode with the Closed Loop Stimulation (CLS) function OFF
  Interventions: Device: DDD(R)

INTERVENTIONS:
Device: DDD+CLS — Device will be programmed in a dual-chamber DDD pacing mode with the Closed Loop Stimulation (CLS) function ON
  Arms: Active group - CLS ON
Device: DDD(R) — Device will be programmed in a dual-chamber DDD(R) pacing mode with the Closed Loop Stimulation (CLS) function OFF
  Arms: Control group - CLS OFF

SUMMARY:
The study is designed as a multi-center, international, prospective, parallel, randomized, single blinded trial comparing the time to first primary endpoint event (Sustained Paroxysmal AF/Persistent AF or stroke/TIA) occurrence in a follow up period of 3 years, between Closed Loop Stimulation (CLS) ON versus OFF, on top of a DDD pacing in patients with pacemaker or ICD indication who require dual-chamber pacing due to sinus node disease (SND), with or without atrioventricular (AV) block.

DETAILED DESCRIPTION:
The benefits of rate-responsiveness on top of dual-chamber pacing still need to be definitively assessed in Sinus Node Dysfunction (SND). Although many rate responsive (RR) sensors have been developed, no large clinical trials evaluated their benefits in terms of clinical endpoints such as clinically relevant atrial fibrillation (AF) and stroke. Electromechanical sensors (piezoelectric accelerometers) have been widely used for their simplicity and overall reliability. However there is some evidence indicating the Closed Loop Stimulation as one of the more efficient and physiological sensors.

Two randomized clinical studies have been conducted so far, showing that in the Brady-Tachy Syndrome the CLS algorithm was associated with a significantly lower overall atrial arrhythmia burden as compared both with a DDDR mode based on a standard accelerometric sensor and an atrial overdrive approach.

Both studies yielded consistent results, albeit with a parallel and intraindividual comparison designs, respectively. The atrial arrhythmic burden is an important but surrogate endpoint, not necessarily related to long-term clinical outcome. The CLS effects on AF (if any) should be investigated in terms of time to first new onset of clinically relevant AF.

In the light of these considerations, it appears interesting to run a large randomized study coherently collecting data on the overall clinical benefit of CLS, primarily in terms of AF and stroke, in a population indicated for pacemaker or ICD and needing dual-chamber pacing due to SND.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Class I or II recommendations for permanent pacing due to SND, with or without AV block according to the current guidelines;
* Patients for whom dual-chamber pacing is indicated or preferred;
* Patients with an optimized and stable antiarrhythmic medical therapy at the time of enrolment;
* Closed Loop Stimulation function was not previously activated;
* No stroke events from implant;
* Patient implanted for the first time;

Exclusion Criteria:

* Permanent AF (PermAF)
* NYHA Class IV Heart Failure
* Stage V kidney dysfunction
* Any indication to Cardiac Resynchronization Therapy (CRT)
* Life expectancy < 1
* Minors
* Pregnant or breast-feeding patients
* Participation in another interventional trial
* Atrial fibrillation ablation (left pulmonary veins) or other cardiac surgery < 3 m

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1390 (Actual)
Dates: Start 2015-09; Primary Completion 2023-03 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
First event of Sustained Paroxysmal AF or Persistent AF or stroke or TIA, whichever comes first. | three years

SECONDARY OUTCOMES:
Sustained Paroxysmal AF (SPAF) | Three years
  Assess the date of each events of SPAF occurred during the follow-up periods
Persistent AF | Three years
  Assess the date of each events of peristent AF occurred during the follow-up periods
Permanent AF | Three years
  Assess the date when AF is declared permanent
Stroke/TIA | Three years
  Assess the date of each events of stroke/TIA occurred during the follow-up periods
Worsening Heart failure Hospitalization (wHF-H) | Three years
  Assess the date of each events of wHF-H occurred during the follow-up periods
All cause mortality | Three years

CONTACTS AND LOCATIONS:
Locations (54):
- China (3):
  - Wuhan Asia Heart Hospital, Wuhan, Jinghan District
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Nangang District
  - Xuanwu Hospital Capital Medical University, Beijing, West City District
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- Max Super Speciality Hospital, New Delhi, India
- Italy (34):
  - Ospedali Riuniti di Ancona, Torrette, Ancona
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti, Bari
  - Ospedale "Bolognini", Seriate, Bergamo
  - Presidio Ospedaliero Ospedale Sant'Anna, San Fermo della Battaglia, Como
  - Ospedale Civile SS. Annunziata, Savigliano, Cuneo
  - Ospedale di Rho, Rho, Italia
  - Ospedale F. Ferrari, Casarano, Lecce
  - Ospedale Maria SS Addolorata, Eboli, Salerno
  - Ospedale Santa Maria della Stella, Orvieto, Terni
  - Ospedale di Conegliano, Conegliano, Treviso
  - Azienda Ospedaliera Policlinico Consorziale, Bari
  - Ospedale Antonio Cardarelli, Campobasso
  - Azienda Ospedaliera di Caserta Sant'Anna e San Sebastiano, Caserta
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Ospedale Santa Maria Nuova, Florence
  - Ospedale Fabrizio Spaziani, Frosinone
  - ASST Valle Olona - Ospedale Sant'Antonio Abate, Gallarate
  - ASST RHODENSE - Ospedale Guido Salvini, Garbagnate
  - Ospedale Ferdinando Veneziale, Isernia
  - Ospedale Vito Fazzi, Lecce
  - Nuovo Ospedale delle Apuane, Massa
  - Ospedale V. Monaldi, Napoli
  - A.O.P. Federico II, Napoli
  - A.O.U Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale S. Maria della Misericordia, Perugia
  - Nuovo Ospedale Santo Stefano, Prato
  - Ospedale "Maria Paternò Arezzo", Ragusa
  - Ospedale Infermi di Rimini, Rimini
  - Policlinico Umberto I, Roma
  - Policlinico Casilino, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - Azienda Ospedaliera "S. Maria" di Terni, Terni
  - Ospedale di Treviso, Treviso
- Hospital Serdang, Kajang, Malaysia
- Singapore (2):
  - National Heart Center Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (6):
  - Sejong General Hospital, Bucheon-si
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Seul National University Bundang Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seul National University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (2):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Result] Puglisi A, Altamura G, Capestro F, Castaldi B, Critelli G, Favale S, Pavia L, Pettinati G. Impact of Closed-Loop Stimulation, overdrive pacing, DDDR pacing mode on atrial tachyarrhythmia burden in Brady-Tachy Syndrome. A randomized study. Eur Heart J. 2003 Nov;24(21):1952-61. doi: 10.1016/j.ehj.2003.08.011. PMID 14585254
- [Result] Puglisi A, Favale S, Scipione P, Melissano D, Pavia L, Ascani F, Elia M, Scaccia A, Sagone A, Castaldi B, Musacchio E, Botto GL; Burden II Study Group. Overdrive versus conventional or closed-loop rate modulation pacing in the prevention of atrial tachyarrhythmias in Brady-Tachy syndrome: on behalf of the Burden II Study Group. Pacing Clin Electrophysiol. 2008 Nov;31(11):1443-55. doi: 10.1111/j.1540-8159.2008.01208.x. PMID 18950302
- [Result] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Result] Russo V, Rago A, Papa AA, Golino P, Calabro R, Russo MG, Nigro G. The effect of dual-chamber closed-loop stimulation on syncope recurrence in healthy patients with tilt-induced vasovagal cardioinhibitory syncope: a prospective, randomised, single-blind, crossover study. Heart. 2013 Nov;99(21):1609-13. doi: 10.1136/heartjnl-2013-303878. Epub 2013 May 30. PMID 23723446
- [Result] de Cock CC, Giudici MC, Twisk JW. Comparison of the haemodynamic effects of right ventricular outflow-tract pacing with right ventricular apex pacing: a quantitative review. Europace. 2003 Jul;5(3):275-8. doi: 10.1016/s1099-5129(03)00031-x. PMID 12842643
- [Result] Lieberman R, Grenz D, Mond HG, Gammage MD. Selective site pacing: defining and reaching the selected site. Pacing Clin Electrophysiol. 2004 Jun;27(6 Pt 2):883-6. doi: 10.1111/j.1540-8159.2004.00551.x. PMID 15189520
- [Result] Lamas GA, Lee KL, Sweeney MO, Silverman R, Leon A, Yee R, Marinchak RA, Flaker G, Schron E, Orav EJ, Hellkamp AS, Greer S, McAnulty J, Ellenbogen K, Ehlert F, Freedman RA, Estes NA 3rd, Greenspon A, Goldman L; Mode Selection Trial in Sinus-Node Dysfunction. Ventricular pacing or dual-chamber pacing for sinus-node dysfunction. N Engl J Med. 2002 Jun 13;346(24):1854-62. doi: 10.1056/NEJMoa013040. PMID 12063369
- [Result] Connolly SJ, Kerr CR, Gent M, Roberts RS, Yusuf S, Gillis AM, Sami MH, Talajic M, Tang AS, Klein GJ, Lau C, Newman DM. Effects of physiologic pacing versus ventricular pacing on the risk of stroke and death due to cardiovascular causes. Canadian Trial of Physiologic Pacing Investigators. N Engl J Med. 2000 May 11;342(19):1385-91. doi: 10.1056/NEJM200005113421902. PMID 10805823
- [Result] Toff WD, Camm AJ, Skehan JD; United Kingdom Pacing and Cardiovascular Events Trial Investigators. Single-chamber versus dual-chamber pacing for high-grade atrioventricular block. N Engl J Med. 2005 Jul 14;353(2):145-55. doi: 10.1056/NEJMoa042283. PMID 16014884